CLINICAL TRIAL: NCT04577976
Title: FreeStyle Libre 2 Flash Glucose Monitoring System Control Phase Study for Pediatric Patients - BG
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-PMS-20194
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: SMBG — Subjects and/or their caregivers will utilize capillary SMBG for managing diabetes for 6 months.

SUMMARY:
This is a prospective, multi-center, non-randomized, single-arm study intended to characterize the safety of self-monitoring of blood glucose (SMBG) when used to manage diabetes in pediatric patients.

DETAILED DESCRIPTION:
Approximately 400 subjects aged 4-17 years and older with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes will be enrolled in the study. Subjects and/or their caregivers will utilize capillary SMBG for managing diabetes for 6 months. Subjects and/or their caregivers will maintain a diary/log book of Adverse Events experienced during the duration of the study. Assessment of Adverse Events will occur via self reporting at each monthly visit and/or phone call.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 4 - 17 years of age.
* Subject must have a diagnosis of type 1 or type 2 diabetes mellitus for at least 3 months prior to enrollment.
* Subject is currently using SMBG for managing their diabetes.
* Subject and/or caregiver must be able to read and understand English.
* In the investigator's opinion, the subject and/or caregiver must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Subject and/or parent or guardian must be willing and able to provide written signed and dated informed consent and assent when appropriate.

Exclusion Criteria:

* Subject has previously used a continuous glucose monitoring system to manage their diabetes within the last six (6) months.
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is known to be pregnant or is attempting to become pregnant at the time of enrollment.
* Subject is on dialysis at the time of enrollment.
* Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff.
* Subject currently is participating in another clinical trial.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric subjects aged 4-17 years and older with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes. At least 50% of the study population will be age 4-12 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Safety of the SMBG devices. The safety of self-monitoring of blood glucose (SMBG) when used to manage diabetes in a pediatric patient population will be characterized: Serious Adverse events | six months
  Rate of Serious Adverse events associated with Hypoglycemia and Hyper glycaemia will be determined. (e.g severe hypoglycemic occurrences requiring health care professional (HCP) intervention including EMT assistance, hospital/clinic visit and/or hospitalization and moderate hypoglycemia in which the patient required the assistance of another person [e.g. as a result of confusion, coma, or seizure] during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (2):
- United States (2):
  - Florida Institute, Orlando, Florida
  - The DOCS, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No